CLINICAL TRIAL: NCT04929977
Title: Evaluation of a m-Health System for Tracking Kangaroo Mother Care and Temperature for Providing Feedback to Family Care Givers or Front-line Workers to Enhance Kangaroo Mother Care Adherence
Brief Title: m-Health System for Tracking Kangaroo Mother Care and Temperature in Southern India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. John's Research Institute (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: OPP1182699
Record Dates: First submitted 2017-12-19; First posted 2021-06-18 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Preterm Infant; Low Birth Weight Infant; Kangaroo Mother Care; Hypothermia, Newborn; Fever
MeSH Terms: conditions — Premature Birth; Hypothermia; Fever | interventions — Wearable Electronic Devices

STUDY DESIGN:
Intervention Model Description: Wearable device combined with a smart mobile phone and back-end analytics system that acts as a temperature and touch sensor and actuator will be evaluated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wearable device with smart mobile phone (Other): 20 mother/care provider-infant pairs practicing Kangaroo Mother Care, from a tertiary super-specialty hospital selected to wear the device ( few days in the hospital and for a week at home when discharged)
  Interventions: Device: Wearable device with smart mobile phone

INTERVENTIONS:
Device: Wearable device with smart mobile phone — The wearable device will act as a sensor designed to identify critical parameters such as Kangaroo Mother Care adherence and temperature of the infant 24/7 and of the mother-infant pairs during these sessions.

SUMMARY:
The product innovation is a wearable device that (combined with a smartphone and back-end analytics system) acts as a sensor, processor and actuator, and is therefore designed to identify critical parameters (Kangaroo Mother Care adherence and temperature of neonate on a 24/7 basis and temperature of mother during these episodes), make intelligent and early diagnosis of (persistent or impending) neonatal hypothermia, maternal/neonatal fever and non-adherence to Kangaroo Mother Care and then trigger audio or visual alerts (via the wearable or smart-mobile phone) for action by the care-giver or front-line healthcare worker to enhance Kangaroo Mother Care duration or referral to a health facility as needed.

DETAILED DESCRIPTION:
Project design and implementation plan:

The logic model envisioned in this study as i) wearable sensors, technology design and development with research team personnel as 'inputs'; ii) data analytics deployment with detection of abnormalities as 'processes'; and iii) feedback alerts appraisal as the 'outputs' for this phase of testing.

Experimental plan comprises of two steps: a non-clinical phase and a clinical phase.

i) The non-clinical phase comprises of the design, development and deployment of the data capture and analytics system. This includes mobile phone app building with features such as push notifications, offline data storage and synchronization on connectivity, local data analysis (with sequentially increasing capabilities as more data comes in) and alerting stakeholders. In addition, capability development of primary nodes for temporary storage and real-time data analysis as also for long-term data storage capabilities that could be scaled to district-level and state-level expansion in future will be done. Data monitoring capacity will be built on real-time visualization dashboards and raising alerts for targeted stakeholders. The entire computational hardware, algorithms/AI engine, network architecture, overall data visualization including heat maps (infrastructure) for this proposed study will be developed by industry experts (will be subcontracted).

ii)In the second phase, it is proposed to undertake a technological-feasibility study as a small-scale clinical trial (in a convenient sample of 20 mother-baby pairs) for testing in real-world conditions while the mother-infant pairs are in the hospital for a few days and when they are discharged for follow-up at home for up to a week. This phase will also include a qualitative research component to study acceptability and feasibility of alerting and actionable advisories sent to care-givers and field staff. All data obtained from this program will reside within dedicated servers with storage facilities within the selected hospital from where mother-infant pairs are recruited. Institutional Ethics Committee approval, clinical trial registration and data safety monitoring board constitution will be undertaken to protect human research participants.

ELIGIBILITY:
Inclusion Criteria:

* Stable LBW babies who are less than 2000 grams
* Kangaroo care provider who could preferably be the mother or any other family member

Exclusion Criteria:

* Extreme preterm infants (corrected gestational age less than 28 weeks)
* Any family member who is unwilling to hold the infant in Kangaroo Mother Care position with the wearable device or if presenting with any infection

Ages: 2 Days to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of hypothermia episodes through the wearable device (remote bio-monitoring - RBM) in real world | 5 months
  1. Number of hypothermia (less than 36.5 degree centigrade) episodes
Evaluation of touch through the wearable device (remote bio-monitoring - RBM) in real world | 5 months
  1. No Kangaroo Mother Care ( Skin to skin contact between mother and baby) for 6 hours (alerted through RBM device)

SECONDARY OUTCOMES:
Development of entire computational hardware of the remote bio-monitoring device | 8 months
  1. No of alert messages from the RBM to project staffs.
  2. No of heat map views - total and within 24 hrs.
  3. No of responses to failure of normal temperature range (36.5-37 degree centigrade/ Kangaroo Mother Care alerts)

CONTACTS AND LOCATIONS:
Overall Officials: Prem K Mony, MD; MSc-Epi, Principal Investigator — St. John's Research Institute, Bangalore 560034
Locations (1):
- St Johns Medical College and Hospital, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Conde-Agudelo A, Diaz-Rossello JL. Kangaroo mother care to reduce morbidity and mortality in low birthweight infants. Cochrane Database Syst Rev. 2014 Apr 22;(4):CD002771. doi: 10.1002/14651858.CD002771.pub3. PMID 24752403
- [Background] Baig MM, Gholamhosseini H, Connolly MJ. A comprehensive survey of wearable and wireless ECG monitoring systems for older adults. Med Biol Eng Comput. 2013 May;51(5):485-95. doi: 10.1007/s11517-012-1021-6. Epub 2013 Jan 19. PMID 23334714
- [Background] Bergh AM, Manu R, Davy K, van Rooyen E, Asare GQ, Williams JK, Dedzo M, Twumasi A, Nang-Beifubah A. Translating research findings into practice--the implementation of kangaroo mother care in Ghana. Implement Sci. 2012 Aug 13;7:75. doi: 10.1186/1748-5908-7-75. PMID 22889113
- [Background] Engmann C, Wall S, Darmstadt G, Valsangkar B, Claeson M; participants of the Istanbul KMC Acceleration Meeting. Consensus on kangaroo mother care acceleration. Lancet. 2013 Nov 30;382(9907):e26-7. doi: 10.1016/S0140-6736(13)62293-X. Epub 2013 Nov 16. No abstract available. PMID 24246562
- [Background] Fink G, Ross R, Hill K. Institutional deliveries weakly associated with improved neonatal survival in developing countries: evidence from 192 Demographic and Health Surveys. Int J Epidemiol. 2015 Dec;44(6):1879-88. doi: 10.1093/ije/dyv115. Epub 2015 Jun 30. PMID 26130739
- [Background] Lawn JE, Kinney MV, Belizan JM, Mason EM, McDougall L, Larson J, Lackritz E, Friberg IK, Howson CP; Born Too Soon Preterm Birth Action Group. Born too soon: accelerating actions for prevention and care of 15 million newborns born too soon. Reprod Health. 2013;10 Suppl 1(Suppl 1):S6. doi: 10.1186/1742-4755-10-S1-S6. Epub 2013 Nov 15. PMID 24625252
- [Background] Lee YG, Jeong WS, Yoon G. Smartphone-based mobile health monitoring. Telemed J E Health. 2012 Oct;18(8):585-90. doi: 10.1089/tmj.2011.0245. PMID 23061640
- [Background] Mony PK, Jayanna K, Bhat S, Rao SV, Crockett M, Avery L, Ramesh BM, Moses S, Blanchard J. Availability of emergency neonatal care in eight districts of Karnataka state, southern India: a cross-sectional study. BMC Health Serv Res. 2015 Oct 6;15:461. doi: 10.1186/s12913-015-1126-3. PMID 26444272
- [Background] Lund C. Medical adhesives in the NICU. Newborn and Infant Nursing Reviews 2014; 14; 14(4):160-165. DOI: 10.1053/j.nainr.2014.10.001
- [Background] Udani RH, Hinduja ARA, Rao SPN, Kabra NS. Role of Kangaroo Mother Care in Preventing Neonatal Morbidity in the Hospital and Community: A review article. Journal of Neonatology, Oct-Dec 2014; 28 (4):29-36.
- [Background] Varkey P, Horne A, Bennet KE. Innovation in health care: a primer. Am J Med Qual. 2008 Sep-Oct;23(5):382-8. doi: 10.1177/1062860608317695. PMID 18820143